CLINICAL TRIAL: NCT05410990
Title: Predictive Value of Eosinophil Indices for Major Cardiovascular Events in Patients With Acute Heart Failure
Brief Title: Eosinophil Indices in Patients With Acute Heart Failure
Status: Completed | Type: Observational
Sponsor: Giresun University (Other)
Responsible Party: Sponsor
Other Study IDs: 05062015
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Acute Heart Failure; Reduced Systolic Function
Keywords: eosinophil indices, acute heart failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mortality, MACE (+): patients with all-cause mortality within the first 6 months of index hospitalization and MACE (major adverse cardiovascular events)
  Interventions: Diagnostic Test: eosinophil and other hematological parameters
- mortality, MACE (-): patients without all-cause mortality within the first 6 months of index hospitalization and MACE (major adverse cardiovascular events)
  Interventions: Diagnostic Test: eosinophil and other hematological parameters

INTERVENTIONS:
Diagnostic Test: eosinophil and other hematological parameters

SUMMARY:
All consecutive patients admitted to the intensive care unit (ICU) with ADHF between January 2017 and December 2021 were enrolled in this retrospective study. All-cause mortality and MACE were assessed with respect to relationships with eosinophil indices, including neutrophil-to-eosinophil ratio (NER), leukocyte-to-eosinophil ratio (LER), eosinophil-to-lymphocyte ratio (ELR), and eosinophil-to-monocyte ratio (EMR).

DETAILED DESCRIPTION:
All consecutive patients admitted to the intensive care unit (ICU) with ADHF and reduced EF between January 2017 and December 2021 were enrolled in this retrospective study. HFrEF was defined as having an LVEF of ≤40%. Demographic data were retrieved from patient charts and the institutional digital database. Patients with an LVEF >40%, NYHA Class I and II subjects, those with advanced liver, kidney diseases or malignancies, patients in whom life expectancy was extremely short and patients with autoimmune, allergic, or infectious diseases that affect the eosinophil indices were not included in the study. The study was approved by the local ethics committee.

Conventional guidelines had been followed for the in-hospital treatment of all patients with ADHF, including loop diuretics, vasodilators, inotropes/vasopressors [9]. Blood tests including complete blood count, blood urea nitrogen and creatinine, electrolytes, liver enzymes, and NT-pro BNP were ordered upon admission to the ICU. All patients underwent transthoracic echocardiography. LVEF was measured with 2-dimensional echocardiography via the modified Simpson method [10]. Data concerning 6-month all-cause mortality and MACE were retrieved from the institutional digital database. The definition of MACE was the composite of total death and re-hospitalization for HF within 6 months of initial hospitalization.

The primary outcome measure of this study was all-cause mortality within the first 6 months of index hospitalization and its relationship with eosinophil indices, including NER, LER, ELR and EMR. The secondary outcome measure of this study was the assessment of MACE within the first 6 months of index hospitalization and its association with eosinophil indices.

ELIGIBILITY:
Inclusion Criteria:

* patients who admitted to the intensive care unit (ICU) with Acute Decompensated Heart Failure and reduced Ejection Fraction (<%40)

Exclusion Criteria:

* Patients with an LVEF >40%, NYHA Class I and II subjects, those with advanced liver, kidney diseases or malignancies, patients in whom life expectancy was extremely short and patients with autoimmune, allergic, or infectious diseases

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acute decompensated heart failure
Sampling Method: Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
mortality | within the first 6 months of index hospitalization
  all-cause mortality

SECONDARY OUTCOMES:
MACE | within the first 6 months of index hospitalization
  major adverse cardiovascular events